CLINICAL TRIAL: NCT01579045
Title: Effect of Head and Gaze Position on Soft Toric Contact Lens Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-005141
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- Sequence 1 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  Filcon II 3, nelfilcon A, etafilcon A, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 2 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  Filcon II 3, nelfilcon A, etafilcon A, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 3 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  Filcon II 3, etafilcon A, nelfilcon A, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 4 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  Filcon II 3, etafilcon A, nelfilcon A, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 5 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  nelfilcon A, Filcon II 3, etafilcon A, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 6 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  nelfilcon A, Filcon II 3, etafilcon A, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 7 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  nelfilcon A, etafilcon A, Filcon II 3, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 8 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  nelfilcon A, etafilcon A, Filcon II 3, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 9 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  etafilcon A, Filcon II 3, nelfilcon A, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 10 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  etafilcon A, Filcon II 3, nelfilcon A, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 11 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  etafilcon A, nelfilcon A, Filcon II 3, senofilcon A, Filcon II 3
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3
- Sequence 12 (Experimental): Five separate sessions of bilateral lens wear of approximately 1 hour. This sequence is as follows:
  etafilcon A, nelfilcon A, Filcon II 3, Filcon II 3, senofilcon A
  Interventions: Device: senofilcon A; Device: etafilcon A; Device: nelfilcon A; Device: Filcon II 3

INTERVENTIONS:
Device: senofilcon A — bilateral daily use soft contact lens
Device: etafilcon A — bilateral daily use soft contact lens
Device: nelfilcon A — bilateral daily use soft contact lens
Device: Filcon II 3 — bilateral daily use soft contact lens
Device: Filcon II 3 — bilateral daily use soft contact lenses

SUMMARY:
Primary Hypotheses:

Senofilcon A will provide significantly less rotation with subjects in a recumbent position than Filcon II 3 monthly .

Etafilcon A will provide significantly less rotation with subjects in a recumbent position than Filcon II 3 1 1 day .

Etafilcon A will provide rotation with subjects a recumbent position non-inferior to nelfilcon A. A margin of 5 degrees will be used.

Secondary Hypotheses:

Senofilcon A will have significantly better monocular visual performance with subjects in a recumbent position than Filcon II 3 monthly.

Etafilcon A for astigmatism will have significantly better monocular visual performance with subjects in a recumbent position than Filcon II 3 1 day.

Etafilcon A will have monocular visual performance with subjects in a recumbent position non-inferior nelfilcon A. A margin of 0.05 LogMAR will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-60 years.
* Read, understand, and sign written Statement of Informed Consent.
* Appear able and willing to adhere to the instructions set forth in the clinical protocol.
* Be existing soft contact lens wearers (no extended wear in the last 3 months, but silicone hydrogels in daily wear are allowed).
* Require a visual correction in both eyes (monovision allowed but no monofit).
* Have a spherical contact lens requirement in the range -1.00 to -6.00D.
* Have astigmatism of between -0.75 and -2.00DC in both eyes.
* Have axes of astigmatism within +/-10° of the following available lens axes: 70°, 90°, 110°, 20°, 180° & 160°, i.e. 60-120, 10-30 and 150-180.
* Monocular distance visual acuity correctable to 6/9 or better in each eye with best sphero-cylindrical refraction.
* Have normal eyes with no evidence of any ocular abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  i) Clear cornea ii) No anterior segment disorder iii) No clinically significant slit lamp findings (i.e. edema, staining, scarring, vascularization, infiltrates or abnormal opacities) iv) No other active ocular disease or recent surgery

Exclusion Criteria:

* Having worn rigid gas permeable (RGP) contact lenses within the last 30 days or polymethyl methacrylate (PMMA) contact lenses within the last 3 months.
* Clinically significant corneal edema, corneal vascularization, corneal staining, tarsal abnormalities, bulbar injection or any other abnormality of the cornea that would contraindicate contact lens wear.
* Extended lens wear in last 3 months.
* Any systemic or topical medications that will in the investigator's opinion affect ocular physiology or contact lens performance.
* Any systemic disease affecting ocular health.
* Abnormal lacrimal secretions.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial.
* Any previous anterior ocular surgery.
* Subjects who are known to have an infectious systemic disease (e.g.,hepatitis, tuberculosis).
* Subjects who are known to have an immunosuppressive disease (e.g., HIV positive).
* Subjects who are known to have diabetes.
* Employees or family members of the Research site, Principal Investigator or study team.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Farnham, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and screened based on the inclusion/exclusion criteria.
Groups:
- All Subjects: All subjects who were enrolled.
Period: Overall Study
Arm/Group | All Subjects
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty-four subjects were screened, enrolled and completed each of the two arms of the study. No subjects were deemed ineligible on screening.
Groups:
- Overall Subjects: All subjects who were enrolled, and completed the study.
Arm/Group | Overall Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: Lens Orientation in Recumbent Position
Description: rotation from zero position also described as absolute value of the rotation.
Time Frame: up to 60 minutes in recumbent position
Population: Subjects analyzed were those enrolled, randomized, and whom completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Groups:
- Senofilcon A (AOfA); Filcon II 3 (Sauflon); Etafilcon A (1DAMfA); Filcon II 3 (C1DT); Nelfilcon A (FDT): As this was a non-dispensing study, the study lenses were worn only during the duration of the visit. Study lenses were marked with a non-toxic marker (e.g. surgical pen) prior to use to aid identification of the lens orientation markers. Each subject wore sequentially the 5 study lenses in a bilateral and random fashion at two different visits.
Arm/Group | Senofilcon A (AOfA) | Filcon II 3 (Sauflon) | Etafilcon A (1DAMfA) | Filcon II 3 (C1DT) | Nelfilcon A (FDT)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
degrees | 15.8 [11.23 to 20.44] | 35.2 [30.62 to 39.79] | 19.4 [14.60 to 24.22] | 29.1 [24.23 to 33.95] | 21.7 [16.86 to 26.48]

2. Secondary Outcome: Monocular Visual Acuity in Recumbent Position
Description: Visual Acuity measured in LogMAR units. High contrast visual acuity (VA) was measured in both eyes using a 3m LogMAR test chart at 2.5m testing distance (subsequently converted).
Time Frame: up to 60 minutes in recumbent position
Population: Analysis is on those who were enrolled, randomized, and whom completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale (LogMAR)
Arm/Group | Senofilcon A (AOfA) | Filcon II 3 (Sauflon) | Etafilcon A (1DAMfA) | Filcon II 3 (C1DT) | Nelfilcon A (FDT)
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
units on a scale (LogMAR) | -0.008 [-0.044 to 0.029] | 0.041 [0.005 to 0.077] | 0.024 [-0.008 to 0.055] | 0.081 [0.049 to 0.114] | -0.013 [-0.045 to 0.019]

ADVERSE EVENTS:
Arm/Group | Senofilcon A (AOfA) | Filcon II 3 (Sauflon) | Etafilcon A (1DAMfA) | Filcon II 3 (C1DT) | Nelfilcon A (FDT)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less